CLINICAL TRIAL: NCT04931537
Title: Screening and Application Research of Early Diabetic Nephropathy Markers Based on Lipidomics.
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Second Affiliated Hospital of Wenzhou Medical University (Other); Lishui Country People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: zhengchao-2
Record Dates: First submitted 2021-06-14; First posted 2021-06-18 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-06

CONDITIONS: Diabetic Nephropathy Type 2; Biomarker
Keywords: Diabetic Nephropathy Type 2; Metabonomics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — Serum, plasma and urine samples were collected for serological and metabolomic studies
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Diabetic nephropathy (DN) is one of the major microvascular complications associated with diabetic patients, and also the major global cause of chronic kidney disease and end-stage renal disease (ESRD). Albuminuria and estimated glomerular filtration rate (eGFR) are currently recognized clinical indicators for early diagnosis of DN, however, the sensitivity and specificity are unsatisfactory. The early identification and treatment of DKD are conducive to lowering the risk of kidney damage by as much as 50%. Therefore, it is particularly critical to find new biomarkers to reflect the potential DKD lesions in the clinical silent period earlier and more accurately. Therefore, this study intends to analyze the differentially expressed lipids in early DKD, T2DM and healthy adults by mass spectrometry, and verify the related results by larger samples, so as to screen out early markers of DKD and achieve the ultimate goal of clinical application.

DETAILED DESCRIPTION:
The present study was a scientific research project concurrently conducted by clinical and laboratory. In term of clinical research, the basic personal data, medical history, physical examination and auxiliary examination results of subjects were mainly recorded. Whereas in term of basic research, the serum, plasma and urine samples of patients were collected for serological and metabonomics research to find new biomarkers.

First, we recruited the patients who met the inclusion criteria. The patients' serum, plasma and urine were collected at baseline after obtaining informed patient consent. Simultaneously, the basic information, anthropometric indicators (including height, weight, waist circumference, hip circumference, blood pressure), past history, family history, menstrual history, birth history, medication history, lifestyle of the patients were registered, and the corresponding laboratory examination and auxiliary examination were carried out according to the diagnostic process. All data and data were entered into the database for later analysis. After the initial diagnosis, the patients were enrolled in the current trial. The patients were followed up annually until the last follow-up visit, and the complete follow-up was conducted for at least 5 years. Each follow-up followed the principles of routine clinical diagnosis and treatment. In addition, the patients' serum, plasma and urine samples were collected once a year during follow-up, and a centralized test of glycosylated hemoglobin was performed once a year.

In this study, the pathogenesis of type 2 diabetic nephropathy was explored through multi-center standardized clinical follow-up; The potential mechanism and possible biomarkers in patients with early renal diseases of type 2 diabetes was explored through prospective long-term follow-up, so as to find novel therapeutic approaches and suitable population.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have signed informed consent.
2. Subjects were 20-80 years old and of either gender.
3. Subjects showed good compliance, and the follow-up data was available for >5 years.

Exclusion Criteria:

1. Meet the 1999 World Health Organization (WHO) diagnostic criteria for T1DM、T2DM;
2. Renal diseases caused by other causes, including primary and secondary;
3. All kinds of acute infections;
4. The expected life expectancy (life expectancy or related diseases) was less than 5 years according to the researcher's judgment.
5. Drug users or drug abusers;
6. Sexually transmitted diseases such as viral hepatitis, AIDS and syphilis, and infectious diseases such as tuberculosis are in an active period;
7. Any situation judged by the researcher that affects enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects were 20-80 years old and of either gender
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Urinary Albumin Creatinine Ratio，UACR | 5years
  Urinary Albumin Creatinine Ratio

CONTACTS AND LOCATIONS:
Overall Officials: Chao Zheng, MD,PhD, Principal Investigator — the Second Affiliated Hospital Zhejiang University Schoolof Medicine; Yikai Zhang, PhD, Study Director — the Second Affiliated Hospital Zhejiang University Schoolof Medicine
Locations (1):
- the Second Affiliated Hospital Zhejiang University Schoolof Medicine, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No